CLINICAL TRIAL: NCT01583985
Title: Strategies for Prescribing Analgesics Comparative Effectiveness (SPACE) Trial
Brief Title: Strategies for Prescribing Analgesics Comparative Effectiveness Trial
Acronym: SPACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 11-125
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2018-11

CONDITIONS: Back Pain; Osteoarthritis
Keywords: opioid analgesics; chronic pain; musculoskeletal pain
MeSH Terms: conditions — Back Pain; Osteoarthritis; Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid-intensive (Active Comparator): Opioid-intensive prescribing strategy
  Interventions: Other: Opioid-intensive prescribing strategy
- Opioid-avoidant (Active Comparator): Opioid-avoidant prescribing strategy
  Interventions: Other: Opioid-avoidant prescribing strategy

INTERVENTIONS:
Other: Opioid-intensive prescribing strategy — The opioid-intensive arm emphasizes early use of strong opioid analgesics. Medications will be individually adjusted according to patient preferences and responses.
  Arms: Opioid-intensive
Other: Opioid-avoidant prescribing strategy — The opioid-avoidant prescribing strategy emphasizes non-opioid medications from several drug classes. Medications will be individually adjusted according to patient preferences and responses.
  Arms: Opioid-avoidant

SUMMARY:
Chronic musculoskeletal pain conditions are among the most prevalent conditions in VA primary care. Over the past two decades, improved clinical attention to pain has been associated with exponentially greater use of long-term opioid therapy for chronic non-cancer pain, both within and outside the VA system. Despite this change in practice, the proper place of opioids in chronic pain management continues to be controversial because research has not demonstrated the long-term safety and effectiveness of opioids for chronic musculoskeletal pain. The Strategies for Prescribing Analgesics Comparative Effectiveness (SPACE) Trial will fill a critical gap in the evidence by comparing effectiveness and harms of two clinically relevant analgesic prescribing strategies-one that emphasizes early use of strong opioids and one that delays and minimizes opioid use-for Veterans with chronic back, hip, or knee pain. SPACE is designed to be highly relevant to clinical decision-making in VA primary care and to produce knowledge that will improve the lives of Veterans living with chronic pain.

DETAILED DESCRIPTION:
Background: Chronic musculoskeletal pain conditions are among the most common problems seen in primary care. As the importance of these conditions for the health of individuals and society has been increasingly recognized, use of long-term opioid therapy for chronic musculoskeletal pain has grown exponentially. Unfortunately, research has not kept pace with this change in prescribing practice. Although evidence supports the ability of opioid analgesics to produce short-term reductions in pain intensity, long-term trials evaluating opioid effectiveness are not available. Evidence for effects of opioids on function and quality of life are limited, but observational data indicate that many patients treated with long-term opioids continue to experience severe pain and functional limitations. Furthermore, the long-term harms of opioids are poorly described in the literature. Preliminary investigations suggest a variety of potential harms related to opioid therapy, but the incidence and severity of these harms have not been well-quantified.

Objectives: The main objective of the Strategies for Prescribing Analgesics Comparative Effectiveness (SPACE) Trial is to compare benefits and harms of two prescribing strategies: 1) an opioid-intensive strategy that uses strong opioids, such as morphine, early in treatment, and 2) an opioid-avoidant strategy that optimizes non-opioid medications while delaying and minimizing opioid use. SPACE will evaluate, over 12 months, 1) effects of opioid-intensive versus opioid-avoidant prescribing strategies on pain-related function and pain intensity and 2) adverse effects of opioid-intensive versus opioid-avoidant prescribing strategies, including adverse medication-related symptoms, clinically important adverse events, and changes in physical and cognitive performance. Secondarily, the investigators will examine effects of the two prescribing strategies on health-related quality of life, pain sensitivity, and aberrant drug-related behaviors. The investigators will also conduct a secondary qualitative analysis to better understand patients' perceptions of their response to the interventions and of the value of intervention components.

Methods: SPACE is a pragmatic randomized clinical trial designed to compare the benefits and harms over 12 months of two clinically-relevant prescribing strategies for chronic musculoskeletal pain. Eligible Veterans will be those seen in primary care for chronic back or lower-extremity (hip or knee) arthritis pain who have moderate-severe pain intensity and interference with function. Those currently receiving chronic daily opioid therapy will be excluded. Participants will be randomized to the opioid-intensive (n=138) or the opioid-avoidant (n=138) arm, with stratification by primary pain location (back or hip/knee). Medications in each arm will be adjusted to target improvement in pain, while considering individual patient preferences and responses. Interventions will be delivered in a care management model using the randomly assigned prescribing strategies, automated symptom monitoring, and a structured decision-making approach to guide medication adjustment. Outcome assessors masked to treatment assignment will conduct interviews to assess patient-reported outcomes at 0, 3, 6, 9, and 12 months and will assess physical performance and cognitive function at 0, 6, and 12 months. For the primary outcome, the Brief Pain Inventory (BPI) Interference scale, the study will have 80% power to detect a 1 point difference between groups, assuming 2-sided alpha=0.05 and 20% attrition. Analysis will use an intent-to-treat approach, including all participants in the arm to which they were originally assigned.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with chronic back or lower extremity osteoarthritis pain with moderate-severe intensity and interference with function despite analgesic therapy.

Exclusion Criteria:

* schizophrenia, bipolar disorder, or other psychosis;
* moderately severe cognitive impairment;
* anticipated back, knee, or hip surgery within 12 months;
* anticipated life expectancy of less than 12 months;
* current chronic daily opioid therapy;
* absolute contraindications to either prescribing strategy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin E. Krebs, MD MPH, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Krebs EE, Jensen AC, Nugent S, DeRonne B, Rutks I, Leverty D, Gravely A, Noorbaloochi S, Bair MJ, Kroenke K. Design, recruitment outcomes, and sample characteristics of the Strategies for Prescribing Analgesics Comparative Effectiveness (SPACE) trial. Contemp Clin Trials. 2017 Nov;62:130-139. doi: 10.1016/j.cct.2017.09.003. Epub 2017 Sep 8. PMID 28893675
- [Result] Matthias MS, Donaldson MT, Jensen AC, Krebs EE. "I Was a Little Surprised": Qualitative Insights From Patients Enrolled in a 12-Month Trial Comparing Opioids With Nonopioid Medications for Chronic Musculoskeletal Pain. J Pain. 2018 Sep;19(9):1082-1090. doi: 10.1016/j.jpain.2018.04.008. Epub 2018 Apr 30. PMID 29715520
- [Derived] Kroenke K, Stump TE, Kean J, Krebs EE, Damush TM, Bair MJ, Monahan PO. Diagnostic operating characteristics of PROMIS scales in screening for depression. J Psychosom Res. 2021 Aug;147:110532. doi: 10.1016/j.jpsychores.2021.110532. Epub 2021 May 25. PMID 34052655
- [Derived] Kroenke K, Stump TE, Chen CX, Kean J, Damush TM, Bair MJ, Krebs EE, Monahan PO. Responsiveness of PROMIS and Patient Health Questionnaire (PHQ) Depression Scales in three clinical trials. Health Qual Life Outcomes. 2021 Feb 4;19(1):41. doi: 10.1186/s12955-021-01674-3. PMID 33541362
- [Derived] Kroenke K, Stump TE, Chen CX, Kean J, Bair MJ, Damush TM, Krebs EE, Monahan PO. Minimally important differences and severity thresholds are estimated for the PROMIS depression scales from three randomized clinical trials. J Affect Disord. 2020 Apr 1;266:100-108. doi: 10.1016/j.jad.2020.01.101. Epub 2020 Jan 23. PMID 32056864
- [Derived] Koffel E, Kats AM, Kroenke K, Bair MJ, Gravely A, DeRonne B, Donaldson MT, Goldsmith ES, Noorbaloochi S, Krebs EE. Sleep Disturbance Predicts Less Improvement in Pain Outcomes: Secondary Analysis of the SPACE Randomized Clinical Trial. Pain Med. 2020 Jun 1;21(6):1162-1167. doi: 10.1093/pm/pnz221. PMID 31529104
- [Derived] Krebs EE, Gravely A, Nugent S, Jensen AC, DeRonne B, Goldsmith ES, Kroenke K, Bair MJ, Noorbaloochi S. Effect of Opioid vs Nonopioid Medications on Pain-Related Function in Patients With Chronic Back Pain or Hip or Knee Osteoarthritis Pain: The SPACE Randomized Clinical Trial. JAMA. 2018 Mar 6;319(9):872-882. doi: 10.1001/jama.2018.0899. PMID 29509867

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 25 patients withdrew prior to randomization. 10 were excluded by the study team and 15 declined to be randomized.
Groups:
- Opioid: The opioid prescribing strategy included 3 levels of opioid analgesics. Medications were individually adjusted according to patient preferences and responses.
- Non-opioid: The non-opioid prescribing strategy included 3 levels of non-opioid medications from several drug classes. Medications were individually adjusted according to patient preferences and responses.
Period: Overall Study
Arm/Group | Opioid | Non-opioid
Started | 120 | 120
Included in Primary Analysis (Provided patient-reported outcomes at least one post-randomization follow-up timepoint) | 119 | 119
Completed (Main patient-reported outcomes at 12 months) | 117 | 117
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid | Non-opioid | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 64 | 136
  >=65 years | 48 | 56 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (13.3) | 59.7 (14.0) | 58.3 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 84 | 84 | 168
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 105 | 102 | 207
  Black | 7 | 11 | 18
  Other or Multiple | 7 | 6 | 13
  Missing | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 120 | 120 | 240
Brief Pain Inventory Interference [Mean (Standard Deviation); unit: units on a scale] — range 0-10; higher score is worse
  units on a scale | 5.4 (1.5) | 5.5 (2.0) | 5.5 (1.9)
Brief Pain Inventory Severity [Mean (Standard Deviation); unit: units on a scale] — range 0-10; higher score is worse
  units on a scale | 5.4 (1.5) | 5.4 (1.2) | 5.4 (1.4)
Primary Pain Location [Count of Participants; unit: Participants]
  Back pain | 78 | 78 | 156
  Hip/knee osteoarthritis pain | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory Interference Scale
Description: Measure of pain-related functional interference (range 0-10; higher score is worse)
Time Frame: 3 months, 6 months, 9 months, and 12 months
Population: Patients with at least one follow-up outcome assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Opioid | Non-opioid
Number analyzed (Participants) | 119 | 119
units on a scale
  3 months: number analyzed (Participants) | 106 | 115
  3 months | 3.7 (2.1) | 3.7 (2.2)
  6 months: number analyzed (Participants) | 116 | 116
  6 months | 3.4 (2.1) | 3.6 (2.4)
  9 months: number analyzed (Participants) | 108 | 107
  9 months | 3.6 (2.2) | 3.3 (2.4)
  12 months: number analyzed (Participants) | 117 | 117
  12 months | 3.4 (2.5) | 3.3 (2.6)

2. Secondary Outcome: Brief Pain Inventory Severity Scale
Description: Measure of pain intensity (range 0-10; higher score is worse)
Time Frame: 3 months, 6 months, 9 months, and 12 months
Population: patients with at least one follow-up assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Opioid | Non-opioid
Number analyzed (Participants) | 119 | 119
units on a scale
  3 months: number analyzed (Participants) | 106 | 115
  3 months | 4.3 (1.8) | 4.0 (1.7)
  6 months: number analyzed (Participants) | 116 | 116
  6 months | 4.1 (1.8) | 4.1 (1.9)
  9 months: number analyzed (Participants) | 108 | 107
  9 months | 4.2 (1.7) | 3.6 (1.7)
  12 months: number analyzed (Participants) | 117 | 117
  12 months | 4.0 (2.0) | 3.5 (1.9)

3. Secondary Outcome: Medication-related Symptom Checklist
Description: Checklist of bothersome medication-related symptoms (0-19, higher number = more symptoms)
Time Frame: 3 months, 6 months, 9 months, and 12 months
Population: those with any follow-up outcomes
Measure: Mean (Standard Deviation); unit: symptoms
Arm/Group | Opioid | Non-opioid
Number analyzed (Participants) | 119 | 119
symptoms
  3 months: number analyzed (Participants) | 106 | 114
  3 months | 2.3 (2.5) | 1.3 (1.8)
  6 months: number analyzed (Participants) | 115 | 115
  6 months | 2.1 (2.7) | 1.3 (2.3)
  9 months: number analyzed (Participants) | 108 | 107
  9 months | 1.9 (2.8) | 0.9 (1.9)
  12 months: number analyzed (Participants) | 114 | 114
  12 months | 1.8 (2.6) | 0.9 (1.8)

4. Secondary Outcome: Falls
Description: Number of falls in 12 months after enrollment
Time Frame: 12 months
Population: Patients reporting falls at any outcome timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid | Non-opioid
Number analyzed (Participants) | 118 | 119
Participants
  No falls | 63 | 63
  1 fall | 26 | 17
  2 or more falls | 29 | 39

5. Secondary Outcome: Hospitalizations
Description: All cause, EMR-confirmed hospitalizations
Time Frame: 12 months
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid | Non-opioid
Number analyzed (Participants) | 120 | 120
Participants
  No hospitalizations | 99 | 99
  1 hospitalization | 15 | 16
  2 or more hospitalizations | 6 | 5

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Opioid | Non-opioid
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/120
Serious Adverse Events (participants affected / at risk) | 19/120 | 22/120
Other Adverse Events (participants affected / at risk) | 58/120 | 49/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opioid (N=120) | Non-opioid (N=120)
Hospitalization (General disorders) | 19 (23) | 22 (26) — All-cause hospitalizations
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opioid (N=120) | Non-opioid (N=120)
Emergency Department visits (General disorders) | 58 (110) | 49 (81) — All cause ED visits

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2012-05-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT01583985/Prot_000.pdf
  • Statistical Analysis Plan (2011-12-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT01583985/SAP_001.pdf